CLINICAL TRIAL: NCT01947348
Title: Safety and Clinical Effectiveness of A3 SVF in Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Regenerative and Cellular Medicine (Industry)
Responsible Party: Principal Investigator, barbara krutchkoff, Dr John Huh, Los Angeles, Institute of Regenerative and Cellular Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3-912-OA-801
Record Dates: First submitted 2013-03-15; First posted 2013-09-20 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Therapeutics; Cell Extracts

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment with A3 SVF (Experimental): These patients that have been treated. The control patients that have not been treated.
  Interventions: Procedure: treatment with A3 SVF

INTERVENTIONS:
Procedure: treatment with A3 SVF — Treatment interarticular and IV with A3 SVF
  Other Names: A3 SVF, Cell Extracts, Adipose Derived Stem Cells

SUMMARY:
To purpose of this study is to determine if treatment with SVF (Stromal Vascular Fraction) has an effect on pain and inflammation associated with Osteoarthritis.

DETAILED DESCRIPTION:
This is a prospective non-randomized, clinical study of 30 patients to determine safety and treatment potential of A3(Adult Autologous Adipose) SVF for the pain and inflammation associated with Osteoarthritis.

Patients will be treated for Osteoarthritis due to degeneration or chronic injury. They will be given autologous SVF extract derived by the A3 method mixed with activated platelets from a PRP(platelet rich plasma) preparation as direct injections to the effected joints. Outcomes will be tracked with WOMAC (Western Ontario and McMaster Universities Arthritis Index), AUSCAN(Australian Hand Osteoarthritis Index) scores, and a general blood panel in order to evaluate systemic effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication of Osteoarthritis. Can be from degeneration or chronic injury.
* Patients range from 15-90 years of age.
* Female patients not pregnant or lactating.
* Patients with a history of or current corticosteroid therapy will only be eligible if use is suspended from 1 month prior to cell therapy.
* Patients must be able to comply with treatment plan, laboratory tests and periodic interviews.
* Patients with adequate renal function, creatinine ≤ 1.5 mg/dl.
* Patients with adequate blood coagulation activity, PT(INR) < 1.5, APTT <1.5×control.

Exclusion Criteria:

* Diagnosis of cancer within 5 years prior to screening, except for cutaneous basal cell or squamous cell cancer resolved by excision.
* Signs and symptoms of clinically significant cardiac disease.
* Diagnosis of a transient ischemic attack in the 6 months prior to screening,
* Known allergy to anesthetic or any other components of study.
* Patients infected with hepatitis B, C or HIV.
* Patients with Body Mass Index (BMI) > 39kg/m2 .
* Any other cardiovascular illness that in the opinion of the investigator would render a patient unsuitable to participate in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Pain and Inflammation - WOMAC scores, comprehensive inflammation blood panel | one year

SECONDARY OUTCOMES:
Pain and Mobility Assessment | one year

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Krutchkoff, Study Chair — Institute of Regenerative and Cellular Medicine; John Huh, MD, Principal Investigator — ICMS
Locations (1):
- Dr John Huh, Los Angeles, California, United States

REFERENCES:
- See also: IRB — http://www.cellmedicinesociety.org/
- See also: Info regarding outcome measures — http://www.auscan.org/womac/index.htm